CLINICAL TRIAL: NCT01761656
Title: Atorvastatin for Reduction of Myocardial Damage During Angiography and Its Mechanism Associated With IMR
Acronym: ARMYDA-IMR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Zhishan SUN, Central South university, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ARMYDA-IMR 01
Record Dates: First submitted 2012-12-28; First posted 2013-01-07 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Stable Angina; Unstable Angina; Acute Non-ST-segment Elevation Myocardial Infarction
Keywords: stable angina; unstable angina; acute non-ST-segment elevation myocardial infarction; PCI; perioperative myocardial infarction; major adverse cardiac events
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction; Cardiovascular Diseases | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- loading dose atorvastatin (Experimental): For the arm of loading dose atorvastatin, patients will be treated with 80 mg atorvastatin 12 hours before PCI and 40 mg atorvastatin 2 hours before PCI and then 20mg/d after PCI.
  Interventions: Drug: loading dose atorvastatin
- conventional dose atorvastatin (Active Comparator): For the arm of conventional dose atorvastatin, patients will be treated with 20 mg atorvastatin 12 hours before PCI and then 20mg/d after PCI.
  Interventions: Drug: conventional dose atorvastatin

INTERVENTIONS:
Drug: loading dose atorvastatin — For loading dose atorvastatin intervention, patients will be treated with 80 mg atorvastatin (lipitor) 12 hours before PCI and 40 mg atorvastatin (lipitor) 2 hours before PCI and then 20mg/d after PCI.
  Other Names: lipitor
  Arms: loading dose atorvastatin
Drug: conventional dose atorvastatin — For conventional dose atorvastatin intervention, patients will be treated with 20 mg atorvastatin (lipitor) 12 hours before PCI and then 20mg/d after PCI.
  Other Names: lipitor
  Arms: conventional dose atorvastatin

SUMMARY:
The purpose of this study is to determine whether preoperative loading dose atorvastatin can prevent perioperative myocardial infarction during angiography and main adverse cardiac events 1 month after operation in stable angina, unstable angina and acute non-ST-segment elevation myocardial infarction patients undergoing elective coronary angiography and PCI, and determine whether its mechanisms are associated with microcirculation resistance.

DETAILED DESCRIPTION:
With 20 years of popularity of the clinical applications of percutaneous coronary intervention (PCI), increasing attention has been paid to postoperative myocardial injury (MI) after PCI. NAPLES II1 and ARMYDA2Studies have shown that loading dose statin therapy before PCI for ACS patients can reduce perioperative myocardial infarction and major adverse cardiac events (MACE) and mortality 1 year after PCI. The core mechanism about the effects of statins on the clinical outcomes above-mentioned, which can not been completely explained by the lipid-lowering effect, so far have not been discovered in previous studies. Thus the interest of some researchers turned to the other point of view, such as coronary microcirculation. MI after PCI is a kind of non-ST-segment elevation myocardial infarction (NSTEMI) related to coronary microcirculation, which can not been detected by coronary angiography, but can be detected by index of microcirculatory resistance (IMR) examination.

In this study, we will recruit stable angina, unstable angina and acute non-ST-segment elevation myocardial infarction patients who have been confirmed by coronary angiography. At the time of enrollment, patients will be randomly assigned to loading dose group (atorvastatin 80 mg 12 hours before PCI and 40 mg 2 hours before PCI and then 20mg/d after PCI) or control group (atorvastatin 20 mg 12 hours before PCI and then 20mg/d after PCI). When PCI is performed, index of microvascular resistance (IMR) will be measured before and after the procedure. Periprocedural myocardial infarction will be defined by post-PCI cardiac biomarker. All patients will be followed for adverse cardiac events for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina
* Patients with unstable angina patients
* Patients with acute non STsegment elevation myocardial infarction
* Patients willing to accept the need regular follow-up of this study
* Patients 18-75 years of age
* Patients who signed an informed consent form

Exclusion Criteria:

* ST segment elevation acute myocardial infarction
* Emergency coronary angiography in patients
* Patients with abnormal liver function
* Heavily calcified, distortions coronary lesions
* LVEF <30% of patients
* eGFR<30ml/min/1.73 Square meters
* Liver disease or a history of muscle disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
perioperative myocardial infarction | 1 month after PCI

SECONDARY OUTCOMES:
major adverse cardiac events (MACE) 1 month after PCI | 1 month
mortality 1 month after PCI | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Zhishan SUN, doctor, Study Chair — Central South University
Locations (1):
- Xiangtan Clinical College affiliated to Central South University, Xiangtan, Hunan, China